CLINICAL TRIAL: NCT05232565
Title: Prospective Multicenter Study to Characterize the REAL-WORLD EVIDENCE Regarding Safety and Performance of the PTCA Catheters Family
Status: Completed | Type: Observational
Sponsor: Arthesys (Industry)
Responsible Party: Sponsor
Other Study IDs: ART-PTCA-01
Record Dates: First submitted 2022-01-31; First posted 2022-02-10 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Coronary Artery Stenosis
MeSH Terms: conditions — Coronary Stenosis | interventions — Angioplasty, Balloon, Coronary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Percutaneous Transluminal Coronary Angioplasty — Angioplasty intervention of coronary vessels or coronary bypass graft stenosis

SUMMARY:
The purpose of this Post market Study is to collect clinical data of the Arthesys PTCA catheters family during angioplasty intervention of coronary vessels or coronary bypass graft stenosis to support MDR submission.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a Percutaneous intervention to a native coronary or coronary bypass graft indication
* Patient >18 years
* Patient who understands the trial requirements and the treatment procedures and provides written informed consent

Exclusion Criteria:

- Patients will not be included if they are under judicial protection, guardianship or curatorship or if they are deprived of their liberty by judicial or administrative decision.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing PTCA procedure
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-07-29 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Efficacy endpoint | Up to end of PTCA procedure
  Balloon successfully reaching and crossing target location, successful inflation, deflation, and retrieval in the guiding catheter
Safety endpoint | Up to end of PTCA procedure
  Successful balloon dilatation without device related adverse event during the dilatation procedure

SECONDARY OUTCOMES:
Performance - pre-dilatation | Up to end of PTCA procedure
  Residual stenosis < 50% and TIMI flow grade 3
Performance - post-dilatation | Up to end of PTCA procedure
  Angiographic success of the device defined as <30% residual stenosis after angiography

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Saint Louis, La Rochelle, France